CLINICAL TRIAL: NCT00185237
Title: A Multicenter, Double-blind, Randomized, Placebo Controlled Study on the Effect of Ultra-low Dose Transdermal Estradiol (Menostar®) on the Incidence and Severity of Hot Flushes, Other Menopausal Symptoms and on Well-being in Postmenopausal Asian Women Over 12 Weeks.
Brief Title: Treatment of Hot Flushes in Asian Women With Ultra-low Dose Estradiol Patch
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91441; 309120
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Hot Flashes
Keywords: Menopause
MeSH Terms: conditions — Hot Flashes | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Menostar (estradiol transdermal delivery system)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Menostar (estradiol transdermal delivery system) — Menostar (estradiol transdermal delivery system (SHP00577E), 0.014 mg/day)
  Arms: Arm 1
Drug: Placebo — Placebo patch
  Arms: Arm 2

SUMMARY:
150 postmenopausal Asian women with vasomotor symptoms, after fulfilling the inclusion and exclusion criteria will be enrolled in the study. The women will be randomly assigned to one of two treatment groups (Menostar® or placebo), after which they will be asked to use a patch once a week for 12 weeks.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of postmenopausal status

Exclusion Criteria:

* Contraindication to estrogen therapy

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2005-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Relative change in frequency of hot flushes | 12 weeks

SECONDARY OUTCOMES:
Change in intensity of hot flushes | 12 weeks
Changes in vaginal pH | 12 weeks
Changes in vaginal maturation index | 12 weeks
Occurrence of urogenital symptoms | 12 weeks
Change in MENQOL (menopausal quality of life questionaire) | 12 weeks
Bleeding profile | 12 weeks
Safety | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer